CLINICAL TRIAL: NCT02078245
Title: Quality Control Study of MR Based Screening of Individual With Increased Risk for Pancreas Cancer
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Karolinska University Hospital (Other)
Responsible Party: Principal Investigator, Matthias Löhr, Professor, Karolinska University Hospital
Other Study IDs: 2010/1001-32; 2010/1001-32 (Other: Swedish Ethical Board Karolinska Institutet)
Record Dates: First submitted 2014-02-14; First posted 2014-03-05 (Estimated); Last update posted 2023-10-24 (Actual); Status verified 2023-10

CONDITIONS: Hereditary Pancreatitis; Hereditary Pancreatic Cancer
Keywords: Familial pancreatic cancer; Surveillance; Screening
MeSH Terms: conditions — Hereditary pancreatitis; Pancreatic carcinoma, familial

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 15 Years
Biospecimen Retention: Samples With DNA — Bloodsamples
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Familial pancreatic cancer patients: Individual with ten fold higher risk to develop pancreatic cancer.
  Interventions: Other: MRI

INTERVENTIONS:
Other: MRI — MRI

SUMMARY:
Early detection of pre-cancerous lesions or early stage pancreatic cancer seems to have a positive impact in survival for patients with an increased genetic risk to develop pancreas cancer.

In this study, following the indication of the swedish guidelines, consecutive patients with a family history for pancreas cancer underwent a clinical surveillance Magnetic Resonance Imaging (MRI) based. The results of this study were analyzed looking in the patients files collected during the screening period.

DETAILED DESCRIPTION:
Pancreatic cancer is the 4th cause of cancer related deaths in USA and in many of the Western Countries. The incidence of the disease is almost corresponding to the mortality rate. For this reason pancreatic cancer can be considered a global lethal disease. Even if treatments have improved, the resection rate in patients suffering from ductal adenocarcinoma remain around 30% and the 5 years survival rates is below 20%. Because of the low incidence of pancreatic cancer in the general population, a population-based screening is not cost/effective. Anyway in the last two decades, data from literature demonstrate that pancreatic cancer can be the phenotypic expression of some know genetic syndromes and the existence of a familial risk to develop pancreatic cancer. In particular for this last condition, called familial pancreatic cancer (FPC), an increased risk is associated with the number of family member affected. In prospective epidemiological studies, is demonstrated that a positive family history of pancreatic cancer is present in about 10% of all consecutive probands. The identification of a population at risk, the suggestions that an early surgical treatment of pancreatic cancer can improve the prognosis and, in particular, the identifications of pre-neoplastic lesions as PanIN and IPMN associated to the natural history of FPC, contributed to the development on National and International guidelines for the surveillance of the individual at increased risk. Even do, today, no consensus is reached on inclusion criteria for a clinical surveillance program, screening modalities and target lesions. Traditionally individual with a 10 fold relative risk to develop pancreatic cancer were considered suitable for a screening program. However, more recently, the CAPS group suggested to include in a surveillance program individuals with a 5 fold higher relative risk. Early pancreatic cancer, IPMN and PanIN lesions are considered the target lesions of a clinical screening, however the concrete possibility to detect PanIN lesions during a surveillance program remain debatable and uncertain.The imaging modality technique used in the existing programs are, alone or in combination, magnetic resonance (MR), computed tomography (CT), endoscopic ultrasound (EUS), endoscopic retrograde cholagiopancreatography (ERCP). Anyway a tendency to use low aggressive modalities as MR and EUS is emerging by the recent recommendations. The results of the clinical studies are quite uncertain and difficult to compare due to different screening modalities and inclusion criteria. The yield of FPC screening programs published in literature range from 50 to 1.3%. The cost/effectiveness of a surveillance program for FPC is not already demonstrated.

The aim of this study is to analyze the preliminary result of a prospective clinical surveillance program for individuals at risk for pancreatic cancer using a low aggressive, MR based, screening.

Patients enrollment Patients with an increased "genetic" risk to develop pancreatic cancer will be enrolled in a MR surveillance program at Karolinska University Hospital.

The patients were enrolled in the study from 3 different ways: relative of probands treated for pancreas cancer at karolinska University Hospital and with a positive family history of pancreatic cancer or with a positive anamnesis of an associated genetic syndrome, subjects, with a "genetically" increased risk, referred to us from other swedish centers, subjects referred to us by general partitioners.

Inclusion criteria for the screening All the individuals with a 10 fold higher relative risk in respect to the general population to develop pancreatic cancer will be included in the study. In case of suspected known genetic syndromes, only patients with detected corresponding gene mutations will be enrolled.

Screening modalities All patients fulfilling the inclusion criteria will be enrolled in the clinical study after a specific informed consent. Basically a complete familial and personal anamensis (including the pedegree) and a clinical examination will be obtained from all the patients. A blood sample will be collected into a bio-bank at Karolinska University Hospital. An MR/MRCP with secretin will be performed for all the patients. If the result of the MR are negative (no findings detected) a one year screening, with the same modalities is recommended. Only patients with some anomaly at the MR will undergo EUS with or without FNA and/or MDCT scan. Patients with a positive anamnesis suggestive for a known genetic syndrome will be offered specific genetic tests (BRCA1/2, SPINK1, PRSS1, p16, STK11) and respective genetic counselling.

Target lesions of the screening Due to the low specificity and sensibility of the available technique in order to detect PanIN lesions, the lobulocentric atrophy areas are not considered a target of our screening. Macroscopic pre-neoplastic lesions (IPMN) or pancreatic solid mass are considered the only lesions suitable for detection and screening.

ELIGIBILITY:
Inclusion Criteria:

* 10 fold higher risk to develop pancreatic cancer
* Obtained informed consent

Exclusion Criteria:

* age less than 18 yrs
* No consensus obtained

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Familial risk for pancreatic cancer
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2010-08 (Actual); Primary Completion 2025-01 (Estimated); Study Completion 2025-01 (Estimated)

PRIMARY OUTCOMES:
MRI accuracy | Three years
  MRI accuracy in detection precancerous pancreatic lesions.

SECONDARY OUTCOMES:
Definition of spectrum of precancerous pancreatic lesions | During three years
Outcome of surveillance program | Three years
  Outcome of surveillance program analysis

CONTACTS AND LOCATIONS:
Overall Officials: Marco del Chiaro, ass. prof., Principal Investigator — Karolinska University Hospital
Locations (1):
- Gastrocentrum Karolinska University Hospital, Stockholm, Sweden

REFERENCES:
- [Background] Canto MI, Harinck F, Hruban RH, Offerhaus GJ, Poley JW, Kamel I, Nio Y, Schulick RS, Bassi C, Kluijt I, Levy MJ, Chak A, Fockens P, Goggins M, Bruno M; International Cancer of Pancreas Screening (CAPS) Consortium. International Cancer of the Pancreas Screening (CAPS) Consortium summit on the management of patients with increased risk for familial pancreatic cancer. Gut. 2013 Mar;62(3):339-47. doi: 10.1136/gutjnl-2012-303108. Epub 2012 Nov 7. PMID 23135763
- [Background] Bartsch DK, Dietzel K, Bargello M, Matthaei E, Kloeppel G, Esposito I, Heverhagen JT, Gress TM, Slater EP, Langer P. Multiple small "imaging" branch-duct type intraductal papillary mucinous neoplasms (IPMNs) in familial pancreatic cancer: indicator for concomitant high grade pancreatic intraepithelial neoplasia? Fam Cancer. 2013 Mar;12(1):89-96. doi: 10.1007/s10689-012-9582-y. PMID 23179793
- [Result] Pozzi Mucelli RM, Moro CF, Del Chiaro M, Valente R, Blomqvist L, Papanikolaou N, Lohr JM, Kartalis N. Branch-duct intraductal papillary mucinous neoplasm (IPMN): Are cyst volumetry and other novel imaging features able to improve malignancy prediction compared to well-established resection criteria? Eur Radiol. 2022 Aug;32(8):5144-5155. doi: 10.1007/s00330-022-08650-5. Epub 2022 Mar 11. PMID 35275259
- [Result] Del Chiaro M, Ateeb Z, Hansson MR, Rangelova E, Segersvard R, Kartalis N, Ansorge C, Lohr MJ, Arnelo U, Verbeke C. Survival Analysis and Risk for Progression of Intraductal Papillary Mucinous Neoplasia of the Pancreas (IPMN) Under Surveillance: A Single-Institution Experience. Ann Surg Oncol. 2017 Apr;24(4):1120-1126. doi: 10.1245/s10434-016-5661-x. Epub 2016 Nov 7. PMID 27822633
- [Result] Capurso G, Signoretti M, Valente R, Arnelo U, Lohr M, Poley JW, Delle Fave G, Del Chiaro M. Methods and outcomes of screening for pancreatic adenocarcinoma in high-risk individuals. World J Gastrointest Endosc. 2015 Jul 25;7(9):833-42. doi: 10.4253/wjge.v7.i9.833. PMID 26240684
- [Result] Del Chiaro M, Verbeke CS, Kartalis N, Pozzi Mucelli R, Gustafsson P, Hansson J, Haas SL, Segersvard R, Andren-Sandberg A, Lohr JM. Short-term Results of a Magnetic Resonance Imaging-Based Swedish Screening Program for Individuals at Risk for Pancreatic Cancer. JAMA Surg. 2015 Jun;150(6):512-8. doi: 10.1001/jamasurg.2014.3852. PMID 25853369